CLINICAL TRIAL: NCT02240771
Title: Randomized Control Trial of Transarterial Chemotherapy (TAC) Versus Oral Thalidomide and Capecitabine in the Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Transarterial Chemotherapy Compared With Oral Chemotherapy in the Treatment of Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Subrat Kumar Acharya, Professor & Head, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAC-HCC
Record Dates: First submitted 2014-08-31; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Transarterial chemotherapy; Thalidomide; Capecitabine
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transarterial chemotherapy (Active Comparator): Doxorubicin 50mg, Cisplatin 100mg
  Interventions: Procedure: Transarterial chemotherapy
- Oral chemotherapy (Placebo Comparator): Thalidomide---50-300mg once a day Capecitabine---- 500-1500mg once a day
  Interventions: Drug: Oral chemotherapy

INTERVENTIONS:
Procedure: Transarterial chemotherapy — Femoral artery would be punctured at the upper thigh using 18 gauge needle under local anesthesia. Catheterization of the hepatic artery feeding the tumor would be done and placing the catheter tip beyond the gastroduodenal artery, the chemotherapeutic drugs would be administered.
  Mixture would be prepared by using Doxorubicin 50mg and Cisplatin 100mg. Hydrocortisone 100mg and augmenting dose of analgesic and sedative would be injected prior to the administration of the drug.
  The drug mixture would then be injected through the indwelling arterial catheter by continuously flushing alternately, repeatedly and rapidly between two-leur lock syringes.
  Other Names: TAC
  Arms: Transarterial chemotherapy
Drug: Oral chemotherapy — Drugs used would be Thalidomide and Capecitabine in the following dosage schedule- Thalidomide---50mg once a day (OD) for 7 days, increased to 100mg OD for 7 days, 200mgOD for 7 days further increased to 300 mg OD.
  Capecitabine---- 500mg OD for 7 days, then 1000mg OD for next 7 days, increased to a maximum dose of 1500mg OD
  Maintenance dose - Capecitabine 1500 mg - every alternate week Thalidomide - 300 mg OD. Total leucocyte count & Platelet count would be monitored every 15 days
  Other Names: OC
  Arms: Oral chemotherapy

SUMMARY:
In India, majority of our patients have advanced hepatocellular carcinoma (HCC) at presentation and hence are unsuitable for the available curative treatment options. In such patients the treatment options are mainly palliative. Transarterial chemoembolization (TACE), transarterial chemotherapy (TAC) and various forms of oral chemotherapy are the only available options currently. Many patients have more advanced disease with the involvement of branches of portal vein. This further limits the therapeutic options. According to Barcelona Clinic Liver Cancer (BCLC) staging, involvement of portal vein precludes any standard form of therapy. TAC and oral chemotherapy has been tried in this group of patients by few researchers. Which treatment (TAC or oral chemotherapy) would be better suitable for advanced stage (BCLC C) needs to be explored. However, there are no randomized controlled trials (RCT's) available.

TAC is the procedure for treating patients of HCC with portal vein invasion where only the chemotherapeutic drugs are injected into the feeding vessels of the tumor with no subsequent embolization of the feeding vessels.

In order to select a modality which would produce better outcomes in advanced HCC patients (BCLC C), this study was planned.

DETAILED DESCRIPTION:
1. Aim of the study: To see the efficacy of transarterial chemotherapy in prolonging the survival of patients with unresectable HCC when compared to oral chemotherapy 2. Diagnostic criteria

o Cirrhosis of liver- Diagnosis will be founded on the basis of clinical, biochemical, imaging and endoscopy findings.

o Hepatocellular carcinoma- when any one of the following is present

1. Two imaging modalities (dual phase CT (DPCT)/ contrast enhanced MRI) showing arterialization of the hepatic mass
2. Alpha feto protein (AFP) more than 400ng/ml along with arterialization on one imaging modality (DPCT/ contrast enhanced MRI)
3. Fine-needle aspiration cytology (FNAC)

3. Definitions

3.1. Unresectable HCC- • Liver mass larger than 5cm in diameter (single/ multiple) , involving main portal vein with underlying cirrhotic liver

3.2. Tumor response This will be based on Dual phase CT findings

* Complete response (CR)- Tumor fully covered with lipiodol showing no viable tissue
* Partial response (PR)- Tumor partially covered (>75%) by lipiodol
* Mild response (MR)- About 50 to 75% coverage of the tumor by lipiodol
* No response (NR) - About 25 to 50% coverage of the tumor by lipiodol
* Fresh lesions (FL)- Appearance of new mass lesions in the liver with or without recurrence at the site of previous mass

3.3 Patient tolerance Grade 1: no side effects Grade 2: moderate side effects Grade 3: severe side effects Grade 4: life threatening side effects

3.4 Performance status (PST score) PST score of 0-5 would be assessed on the following basis 0- No cancer related symptoms. Normal life style

1. Minor symptoms related to cancer. Capable of non-strenuous activity. Fully ambulatory
2. Ambulatory and capable of all self-care but unable to carry out any work activities. Confined to bed less than 50% of waking hours
3. Capable of only limited self-care. Confined to bed more than 50% of waking hours.
4. Completely disabled. Cannot carry on any self-care. Totally confined to bed.
5. Death

4. Sample Size Systematic review of RCT's for TAC show a 2-year survival of 40 %. Expecting that oral chemotherapy has a 2-year survival of 40% with 5% non-inferiority margin with 80% power and 5% error, a sample size of 124 patients in each arm would be required.(Total 248 patients)

5. Randomization

• Patients will be randomized after the confirmation of diagnosis and obtaining written consent

* Sequences will be generated by the Statistician
* Stratified randomization will be done. Two strata of child's A and B will be made
* Randomization will be done by drawing consecutively numbered opaque sealed envelopes Randomization into A (TAC) and B (oral chemotherapy) will be done

  6. Follow up post TAC

6.1 Clinical follow up

* All patients would be followed up in the Liver clinic monthly unless their clinical condition warrants earlier follow up
* Liver function tests/ complete blood count would also be done at each visit and AFP (if elevated earlier) every six months
* Patient tolerance, child's status would be estimated.

6.2 Imaging follow up

* At one month, a dual phase CT would be done to ascertain the response to therapy and the need to repeat the procedure. Subsequently, the DPCT would be done at 3 and 6 monthly intervals.

  7. Repeat TAC on follow up This would be done if any of the following is noted
* DPCT shows viable tumor
* Fresh lesions appear
* Elevated serum AFP occurs with or without appearance of viable mass on DPCT

ELIGIBILITY:
Inclusion Criteria:

* Patients above 12 years of age with performance status (PST) score of 0-2
* Unresectable HCC with underlying Child's A/B cirrhosis
* Blocked Main portal vein
* No history of drug allergy
* Informed written consent of patient.

Exclusion Criteria:

* Child's C cirrhosis
* Performance status 3-5
* Extra hepatic disease
* Co-morbid illness like coronary artery disease, congestive heart failure, chronic renal failure etc
* Previous history of encephalopathy/ upper gastrointestinal bleed in the last six months
* Pregnancy

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2006-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Survival rate- | 1 year
  Survival rate to be calculated from the start of Transarterial chemotherapy

SECONDARY OUTCOMES:
Tumor response | 1 year
  Tumor response on dual phase contrast-enhanced computed tomography (CECT)

CONTACTS AND LOCATIONS:
Overall Officials: Subrat K Acharya, D.M, Principal Investigator — All India Institute of Medical Sciences, New Delhi, India
Locations (1):
- AII India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India